CLINICAL TRIAL: NCT03897699
Title: Mindful Breathing and Neuromodulation for Depression in Young People
Brief Title: Mindful Breathing and tDCS for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSYCH-2018-26861
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Results first posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Depression; Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Transcranial Direct Current Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- active tDCS + Mindful Breathing Training (Experimental): 20 minutes of active or sham stimulation will be applied at 2.0 mA in parallel with mindful breathing training
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Mindful Breathing
- sham tDCS + Mindful Breathing Training (Sham Comparator): The sham condition will apply stimulation only for the first and last 30 seconds of the 20-minute session
  Interventions: Behavioral: Mindful Breathing; Other: Sham

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — A non-invasive neuromodulation technique that can modulate neural activity. Weak electrical current (~2mA) is applied to the scalp using anodal and cathodal electrode sponges, which increase or decrease cortical excitability respectively.
  Arms: active tDCS + Mindful Breathing Training
Behavioral: Mindful Breathing — MBT is a mindfulness-based intervention that guides participants to pay attention to the present experience. Participants will be trained to become aware of mind-wandering, disengage, and shift attention back to the present experience. Participants will practice mindful breathing using a computerized application that they will be able to access on the web.
Other: Sham — Weak electrical current (~2mA) is applied to the scalp using anodal and cathodal electrode sponges, which increase or decrease cortical excitability respectively. Sham stimulation will serve as a control condition with current applied only for the first and last 30 seconds of the 20-minute session.
  Arms: sham tDCS + Mindful Breathing Training

SUMMARY:
This study will investigate whether transcranial direct current stimulation (tDCS) targeting the dorsolateral prefrontal cortex (DLPFC) can enhance the therapeutic effect of mindful breathing training (MBT) for adolescent depression. The objective is to enhance connectivity between the DLPFC with the amygdala and Default Mode Network (DMN) circuits as well as to enhance emotion regulation abilities and decrease rumination to reduce symptoms of depression. This will aid in the development of novel treatments for depression.

DETAILED DESCRIPTION:
Aim 1: To demonstrate the feasibility of recruiting and randomizing adolescents with depression to a research protocol involving MBT and tDCS. The investigators expect that adolescents will be willing to enroll in a randomized trial involving MBT and tDCS.

Aim 2: To test the tolerability of MBT and tDCS in adolescents. The investigators expect that MBT will be well-tolerated and that active tDCS will show no difference in tolerance compared to sham stimulation.

Aim 3: To examine whether tDCS can enhance the effects of MBT. The investigators expect the MBT + tDCS group will show greater reduction in depressive symptoms compared to the MBT + sham stimulation group.

Aim 4: To examine the mechanisms of MBT +/- tDCS treatment. The investigators expect that depression symptom improvement will be associated with decreased rumination, improvements in emotion regulation, increased task-based and resting state DLPFC-DMN and DLPFC-amygdala connectivity, as well as increased DLPFC activation and reduced amygdala activation during rumination and emotion processing tasks. The investigators also expect reduced alpha asymmetry and reduced LPP amplitude during emotion regulation and emotion processing. The investigators expect these changes will be greatest in the active tDCS + MBT group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder (MDD), Dysthymia, or Other specified/Unspecified Depressive Disorder based on MINI.
* Experiencing current symptoms of depression as indexed by a MADRS-S score ≥ 13
* Ability to access the MBT online-based application (e.g., on a personal laptop, tablet, or cell phone)
* Fluent in English

Exclusion Criteria:

* Any participant with a clinically defined neurological disorder or insult including, but not limited to, a condition likely to increase the risk of seizure; such as, space occupying brain lesion; any history of seizure; history of cerebrovascular accident; transient ischemic attack within two years; cerebral aneurysm; dementia; brain surgery; history or stroke or family history of epilepsy
* Any participant with an increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure or history of significant head trauma with loss of consciousness for ≥ 5 minutes
* Participants with conductive, ferromagnetic, or other magnetic-sensitive metals implanted in the head excluding the mouth that cannot safely be removed. Examples include cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewelry and hair barrettes
* Participants with active or inactive implants (including device leads), including deep brain stimulators, cochlear implants, and vagus nerve stimulators
* Participants with pre-existing sores or lesions at the site of tDCS or EEG electrode placement
* A hair style that would impede EEG and tDCS electrode contact (e.g., dread locks)
* Any participant with a current or possibility of current pregnancy
* Participants unable to give informed consent.
* Participation in any investigational drug trial within 4 weeks of the baseline visit
* Clinically significant laboratory abnormality or medical condition, that in the opinion of the investigator would hinder the participant in completing the procedures required by the study
* Currently actively suicidal with intent and plan determined by the C-SSRS at the baseline visit.
* A diagnosis of current or recent substance use disorder (within the past 12 months)
* A diagnosis of Schizophrenia, Bipolar Disorder, or Autism
* Unstable psychotherapy (therapy must be for at least 3 months prior to entry into the study, with no anticipation of change in the frequency or treatment focus of the therapeutic sessions over the duration of the study)
* Recent change in dose of antidepressant medication (within 6 weeks prior to entry into the study). This includes all antidepressants and any adjunctive psychotropic medications that are being used to address problems related to mood or anxiety (e.g. antipsychotic medications, mood stabilizers)
* Refusal to cooperate with study procedures

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Started | 21 | 22
Completed | 16 | 20
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.2 (2.42) | 20.5 (2.26) | 20.9 (2.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 16 | 27
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in DLPFC Connectivity: Amygdala
Description: Change in dorsolateral prefrontal cortex connectivity with the salience network and the default mode using functional MRI compared between treatment groups: Right Amygdala and left DLPFC. Lower connectivity may represent a reduced tendency to engage in maladaptive, repetitive negative thinking.
  For r-values, 0 represents that the timeseries of the respective ROIs are not correlated. A better outcome may be indexed by lower connectivity (e.g., negative R values), which may represent a greater ability of the DLPFC to downregulate the amygdala and, which in turn may reduce the tendency to engage in maladaptive, repetitive negative thinking.
Time Frame: Baseline and 5 week
Measure: Mean (Standard Deviation); unit: r-value
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Number analyzed (Participants) | 15 | 15
r-value | 0.0977 (0.123) | -0.057 (0.133)

2. Primary Outcome: Change in DLPFC Connectivity: DMN
Description: Change in dorsolateral prefrontal cortex connectivity with the salience network and the default mode using functional MRI compared between treatment groups: default mode network and left DLPFC. Lower DLPFC and DMN connectivity may represent adaptive switching between thinking states to focus on a task at hand or to engage in more reflective, introspective thinking patterns.
  For r-values, 0 represents that the timeseries of the respective ROIs are not correlated. Change in dorsolateral prefrontal cortex connectivity with the salience network and the default mode using functional MRI compared between treatment groups: default mode network and left DLPFC. A better outcome may be indexed by lower DLPFC and DMN connectivity (e.g., negative R values), which may represent adaptive switching between thinking states to focus on a task at hand or to engage in more reflective, introspective thinking patterns.
Time Frame: 5 weeks from baseline
Measure: Mean (Standard Deviation); unit: r-value
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Number analyzed (Participants) | 15 | 15
r-value | 0.0582 (0.139) | -0.00604 (0.106)

3. Secondary Outcome: Change in Depression MADRS-S
Description: Montgomery-Åsberg Depression Rating Scale - self-assessment (MADRS-S) measures change in severity of depression symptoms over time. Treatment response will be measured using the MADRS-S and a ~50% reduction in depression severity, i.e. total MADRS-S score, will indicate a positive response to treatment.
  The scale includes 9 items that are rated by participants on a 4-point Likert scale ranging from 0 - 3. Half-point scores are also possible, i.e 0.5, 1.5, 2.5. Participants rate their symptoms from over the past 3 days and the range of total possible scores is 0 - 27, with a higher score indicating greater severity of symptoms. Bondolfi et al. (2010) found good internal consistency for the MADRS-S, as well as good concurrent validity between the MADRS (clinician administered) and the MADRS-S. Lastly, the MADRS-S was found to be sensitive to change in depression symptoms over time.
Time Frame: Baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Number analyzed (Participants) | 16 | 20
units on a scale | 6.47 (4.69) | 5.95 (4.04)

4. Secondary Outcome: Change in Mindfulness MAAS
Description: Mindful Attention and Awareness Scale (MAAS) measures presence or absence of awareness of what is happening in the present. The MAAS consists of 15 items. Participants are requested to rate each item according to a 6-point Likert scale with the following options: "Almost Always", "Very Frequently", "Somewhat Frequently", "Somewhat Infrequently", "Very Infrequently", and "Almost Never". Previous study reported that the MAAS was internally consistent and a reliable measure. MAAS score ranges from 1 to 6, with a higher score indicating a greater awareness of inner experiences and mindfulness. In the present study, an increase in the total MAAS score would indicate an increase in presence of awareness of what is happening in the present.
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Number analyzed (Participants) | 16 | 20
units on a scale | 0.929 (0.992) | 0.352 (0.859)

5. Secondary Outcome: Change in Rumination RRS
Description: Ruminative Response Scale (RRS) measures rumination, which refers to thoughts and behaviors centered around one's symptoms and their causes, as well as potential consequences. Nolen-Hoeksema, Morrow, & Fredrickson (1993) reported that ruminative thoughts correlated with depressed mood. They further reported a consistency in ruminative responses over a 30-day period. The RRS will be used to measure changes in rumination in the present study. The measure consists of a total of 22 statements that describe ruminative thoughts and participants are requested to rate each statement on a scale of 1 - 4, 1 being "Almost Never" and 4 being "Almost Always". Change in rumination corresponds with a change in the total RRS score.
  Total scores range from 22 to 88.
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Number analyzed (Participants) | 16 | 20
units on a scale | 13.9 (16.6) | 16.1 (12.7)

6. Secondary Outcome: Change in Mindfulness FMI
Description: Freiburg Mindfulness Inventory (FMI) assesses curious attitude toward the mindfulness experience. The FMI contains 14 statements related to mindfulness experiences. Participants are requested to rate each statement according to a 4-point Likert scale ranging from "Rarely" to "Almost Always". An increase in the FMI total score would indicate an increase in mindfulness. Walach et al. (2006) reported that the FMI is a valid and reliable measure of mindfulness.
  Total scores range from 14 to 56.
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: number on a scale
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Number analyzed (Participants) | 16 | 20
number on a scale | 9.07 (8.3) | 6.72 (7.4)

7. Secondary Outcome: Safety: Serious and Non-Serious Adverse Events
Description: Measure of occurrence of negative side-effects from treatment. Side effects will be collected via participant self-report. Number of serious and non-serious adverse events will be considered in determining safety of the treatment. A higher number of adverse events will indicate lower treatment safety.
Time Frame: 9 weeks
Measure: Number; unit: adverse events
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Number analyzed (Participants) | 21 | 22
adverse events | 486 | 654

8. Secondary Outcome: Tolerability: Enrollment and Drop-Out
Description: Number of participants enrolled. A high number of participants enrolled will indicate a higher level of tolerability of the treatment.
Time Frame: 9 weeks
Measure: Number; unit: participants
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Number analyzed (Participants) | 21 | 22
participants | 21 | 22

9. Secondary Outcome: Tolerability: Drop-Out
Description: Number of participants who drop-out due to inability to tolerate treatment. A high number of participant drop-outs will indicate a lower level of tolerability of the treatment.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
Number analyzed (Participants) | 21 | 22
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 9 week period per participant starting at baseline.
Arm/Group | Active tDCS + Mindful Breathing Training | Sham tDCS + Mindful Breathing Training
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 21/21 | 22/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS + Mindful Breathing Training (N=21) | Sham tDCS + Mindful Breathing Training (N=22)
Headache (General disorders) | 10 (21) | 15 (30)
unusual feelings on skin of head (General disorders) | 11 (42) | 17 (88)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (22) | 10 (22)
tingling (General disorders) | 10 (58) | 18 (101)
itchiness (General disorders) | 14 (85) | 21 (152)
sleepliness (General disorders) | 15 (101) | 19 (79)
difficulty paying attention (General disorders) | 11 (40) | 9 (36)
unusual feelings, attitude, emotions (Psychiatric disorders) | 2 (2) | 3 (4)
tooth pain (General disorders) | 1 (1) | 3 (3)
change in hearing (Ear and labyrinth disorders) | 0 (0) | 2 (2)
nausea (Gastrointestinal disorders) | 3 (5) | 4 (8)
twitches (Musculoskeletal and connective tissue disorders) | 4 (9) | 9 (24)
Dizziness (General disorders) | 3 (4) | 6 (9)
anxiety/worry/nervousness (Psychiatric disorders) | 10 (44) | 12 (55)
forgetfulness (General disorders) | 7 (17) | 3 (15)
balance issue (General disorders) | 0 (0) | 2 (2)
hand movement change (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
abnormal sleep (General disorders) | 11 (32) | 9 (24)
muscle knot/ right shoulder stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bike accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT03897699/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03897699/ICF_000.pdf